CLINICAL TRIAL: NCT01806181
Title: Nutrition and Exercise During Adjuvant Treatment (NEXT) Study Implementation of a Physician-referred Exercise and Healthy Eating Intervention as Supportive Care in Breast Cancer Survivors
Brief Title: NEXT (Nutrition and EXercise During Adjuvant Treatment) Study
Acronym: NExT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Kristin Campbell, Kristin Campbell, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H12-02504
Record Dates: First submitted 2013-02-27; First posted 2013-03-07 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cancer Treatment (Other)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
This study will offer a supervised exercise program and healthy eating education to women with breast cancer undergoing chemotherapy as a physician-referred program and measure the adoption, adherence and satisfaction with the intervention as well as its health effects. Past trials have demonstrated various health benefits of exercise yet it is not currently part of supportive care and few suitable programs exist in the community or outside of research. This study is expected to address the unique barriers related to exercise in breast cancer survivors and to better understand how the intervention might work in a real life setting.

DETAILED DESCRIPTION:
HYPOTHESES (Main):

1. The supervised exercise and healthy eating education intervention will be feasible in terms of recruitment (>50%) and retention (>70%) of participants, and; 2) the intervention will be safe and highly acceptable to participants.

JUSTIFICATION: Past trials have demonstrated the benefits of a supervised exercise program in breast cancer survivors during chemotherapy, including reduced side effects of treatment and improvement in physical functioning and quality of life. There are currently no exercise interventions as part of standard cancer care and few suitable programs exist in the community or outside of a research protocol (where they are often associated with strict eligibility criteria and randomization). The proposed study will deliver an exercise and healthy eating program referred by an oncologist as part of supportive cancer care during adjuvant chemotherapy and is expected to specifically address reported barriers to delivery.

OBJECTIVES: The primary aim of this study is to evaluate the feasibility (recruitment rate, adoption and adherence) of a physician referred supervised exercise and healthy eating intervention in newly diagnosed women with breast cancer as supportive care.

The secondary aim is to assess the efficacy for the intervention on:

1. clinical outcomes (chemotherapy completion rate, hospitalization (cancer-related or non-cancer related), and prescriptions written);
2. behaviour change outcomes (steps per day, self-reported physical activity and dietary intake);
3. blood biomarkers of disease recurrence/survival (i.e., IL-6, TNF-α, CRP).

The exploratory aim is to assess patient satisfaction (i.e., program staff, facility, ease of use, parking), healthcare utilization costs (use of medical services and personnel costs related to a cancer diagnosis) and maintenance of lifestyle change (meeting physical activity and healthy eating targets at 1 year post-intervention).

RESEARCH METHOD: This study is a prospective single arm intervention program evaluation study (pre- and post-test design). We aim to recruit women with newly diagnosed early stage curative breast cancer receiving adjuvant chemotherapy over a 12-month period into an exercise and healthy eating program. The intervention will be delivered for the duration of their adjuvant chemotherapy (approximately 12-24 weeks) followed by a 6 month maintenance phase. Women will be referred by their BCCA Vancouver Cancer Centre medical oncologist during their new patient visit or within 1-2 cycles of chemotherapy (see statistical analysis). Participants will be screened for eligibility, and informed consent obtained and a readiness to exercise assessment completed prior to enrollment. The entire intervention is group-based and delivered for the duration of their breast cancer chemotherapy (approximately 12-24 weeks depending on the chemotherapy protocol) followed by a 6 month maintenance phase and one year of non-intervention follow up. The exercise will be a supervised, progressive aerobic and resistance (weight) training program based on past trials and current guidelines, and delivered at a local Breast Cancer Training Centre dedicated exclusively to breast cancer research. The group-based nutrition education session (2-hrs) will be offered at enrollment at the BC Cancer Agency, Vancouver Centre Campus, in addition to 1 hour drop in follow up sessions during the duration of the study. Study outcomes will be measured at baseline, end of chemotherapy, end of maintenance phase and after 12 months of follow up.

STATISTICAL ANALYSIS: Participant characteristics will be summarized using descriptive statistics. The equivalence of participants who were deemed eligible for the intervention compared to all new patients within the same time frame will be assessed in terms of demographic and clinical variables using Student's T-tests for continuous and chi-square tests for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* female;
* aged 19 years and older;
* newly diagnosed with early stage (I-IIIA) breast cancer;
* prescribed adjuvant chemotherapy (with or without radiation) as part of curative treatment for breast cancer; and
* good comprehension of English

Exclusion Criteria:

* contraindications for entry into an exercise program (i.e., known cardiovascular disease, uncontrolled diabetes mellitus, or musculoskeletal impairment issue);
* body mass index (BMI) >40 (morbid obesity);
* mobility impairment requiring use of mobility aids;
* stage IV cancer
* metastatic disease
* neo-adjuvant chemotherapy (with likelihood of surgery after chemotherapy)

Gender exclusion criteria: Male breast cancer is excluded as it is a rare diagnosis.

Age exclusion criteria: Based on enrolling adult participants only. Language exclusion criteria: A good comprehension of English is required to receive instruction on the intervention and complete study forms and evaluations.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-08-06 (Actual); Primary Completion 2016-01-13 (Actual); Study Completion 2016-12-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome will report as recruitment, retention and adherence rates for the sample and their associated 95% confidence intervals | 2 years

SECONDARY OUTCOMES:
Means and standard deviations | 2 years
  The secondary outcomes will be will be summarized with means and standard deviations for normally distributed data and assessed by repeated measures ANOVA to examine change over time

OTHER OUTCOMES:
Healthcare Utilization costs | 2 years
  The exploratory outcomes will be assessed by proportion of participants responses for the patient satisfaction items and healthcare utilization costs will be analyzed by collaborators with the Canadian Centre for Applied Research in Cancer (ARCC).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Campbell, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Breast Cancer Training Center, Vancouver, British Columbia
  - Fitness Centre, Vancouver, British Columbia